CLINICAL TRIAL: NCT07004400
Title: A Blinded Randomized Clinical Investigation of RefluxStop™ Compared With Nissen Fundoplication in the Treatment of Gastroesophageal Reflux Disease (GERD).
Brief Title: A Blinded Randomized Clinical Study of RefluxStop™ Compared With Nissen Fundoplication in the Treatment of GERD
Acronym: RENEW RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Implantica CE Reflux Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RXI005
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: GERD (Gastroesophageal Reflux Disease)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RefluxStop™ device implantation (Active Comparator): Standard surgical technique for implantation RefluxStop™, as described in the Instructions for Use
  Interventions: Device: RefluxStop™ implantation
- Nissen fundoplication surgery (Active Comparator): Standard surgical technique of Nissen fundoplication
  Interventions: Procedure: Nissen fundoplication

INTERVENTIONS:
Device: RefluxStop™ implantation — Standard surgical technique for implantation RefluxStop™, as described in the Instructions for Use
  Arms: RefluxStop™ device implantation
Procedure: Nissen fundoplication — Standard surgical technique for Nissen fundoplication
  Arms: Nissen fundoplication surgery

SUMMARY:
This study will evaluate if the RefluxStop™ device will treat your acid reflux and improve your symptoms and how it compares to the standard surgical treatment for GERD, the Nissen fundoplication.

DETAILED DESCRIPTION:
This study is a post-market prospective, blinded, randomized, multicenter, multi-arm clinical investigation using standard clinical procedures to record data to evaluate the safety and performance of RefluxStop™ compared with standard Nissen fundoplication for the treatment of subjects suffering from GERD.

A randomization will be performed where the Subjects will be blinded as to assigned randomization group.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent and to participate in the clinical investigation;
2. Age ≥ 18 years or according to local legal age of adulthood at the location of the test site if older;
3. Documented GERD present for ≥ 12 months. Typical symptoms are defined as heartburn, which is a burning sensation often presented as a substernal pain;
4. 24-hour pH monitoring proven GERD with pH measurement, off PPI therapy for at least 7 days prior to testing. (Total distal esophageal pH must be < 4 for ≥ 4.5% of time during a 24-hour monitoring);
5. Suitable to undergo general anesthesia and is a suitable laparoscopic surgery candidate as determined by the investigator

Exclusion Criteria:

1. > 8 cm sliding hernia and paraesophageal hernia; no mesh is allowed;
2. Manometry verified lack of or moderate or severe weak peristalsis in esophagus with DCI <300 or pathologic LOS function including hypercontractability, spasm or pathologic nonrelaxing functionality (the latter defined as coordinated swallows in less than 70% of wet swallows or median IRP>15mmHg). Hypercontractability defined as DCI >8'000 or pressure >45 mmHg. Thus, excluding from the study the rare diseases achalasia, scleroderma, and nutcracker esophagus, however, including mild esophageal motility disorder patients with mildly weak peristalsis;
3. History of bariatric or anti-reflux surgery;
4. Female subjects who are pregnant or nursing;
5. Known sensitivity or allergies to silicone materials;
6. Intraoperative findings determined by the investigator that may result in unfavorable conduct of the clinical investigation procedure (as outlined in the IFU);
7. Subjects that are unable to comply with the clinical investigation requirements (for example due to major psychiatric disorder or are considered otherwise unsuitable for participation in the clinical investigation according to the investigator's judgement);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes - Side effects (PROS) evaluation | 6 months
  Patient Reported Outcomes - Side effects (PROS) evaluation at 6 months, combining the well-established side effects of traditional surgical treatment methods:
  * Dysphagia - swallowing difficulties;
  * Odynophagia - pain at swallowing;
  * Inability to belch and inability to vomit; and
  * Worsening of gas bloating compared to baseline;

CONTACTS AND LOCATIONS:
Locations (4):
- Universitätsklinik für Allgemeinchirurgie Klinische Abteilung für Viszeralchirurgie, Vienna, Austria
- Germany (2):
  - St. Elisabethen Krankenhaus Frankfurt, Frankfurt
  - Klinikum Friedrichshafen GmbH, Friedrichshafen
- Klinik Beau-Site Hirslanden Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No